CLINICAL TRIAL: NCT01997047
Title: Improving the Diagnosis of Pediatric Pneumonia at Hospital and Village Levels: A Multi-centre Indian Study
Brief Title: Diagnosing Pneumonia Under Low-resource Conditions
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Seear, Principle Investigator, University of British Columbia
Other Study IDs: H12-00783
Record Dates: First submitted 2013-05-29; First posted 2013-11-27 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Pneumonia; Bronchiolitis; Asthma
Keywords: Pneumonia; bronchiolitis; asthma; children; tachypnea; developing countries; diagnostic criteria
MeSH Terms: conditions — Pneumonia; Bronchiolitis; Asthma; Tachypnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tachypneic children: All tachypneic children under 5 yrs age presenting to study centres. No exclusions.

SUMMARY:
Pneumonia is the commonest cause of death in children worldwide, killing 1.5 million children under the age of 5 years, every year. This is more than the number of children dying from AIDS, malaria and tuberculosis combined. The current diagnostic and management protocols for managing serious respiratory diseases in children are 30 years old and are greatly in need of updating. The successful establishment of useful clinical management criteria for children with respiratory diseases will have benefits for children in low resource regions around the world. The goals of the study are:

* To determine if children with respiratory distress can be reliably diagnosed under low-resource conditions.
* To identify the clinical tests that best differentiate pneumonia from wheezy diseases. These will be used to establish updated diagnostic criteria for common pediatric lung diseases that broaden the current pneumonia algorithm by adding another for wheezy illnesses.
* The ultimate objective is to improve the management and outcome of acute respiratory conditions in children.
* Investigators also wish to test the efficacy of a locally developed cell phone oximeter probe in a low resource setting.

DETAILED DESCRIPTION:
Study organisation. This is a prospective observational study run simultaneously in four Indian public hospitals (King George Medical University, Lucknow; Regency Hospital, Kanpur; Vanivilas Hospital, Bangalore; Bowring and Lady Curzon Hospital, Bangalore). The study started in Oct 2012 to cover the Indian respiratory viral season. In order to maintain high standards of data collection, a post-graduate research coordinator is employed at each hospital. Because of the use of standardised scoring systems and the need for accurate clinical data collection, a member from the Canadian team spent a week at each centre familiarising local research team members with the study protocol and standardised scoring systems. This was followed by a one week trial period of data collection and electronic transmission of files to Canada.

Diagnostic definitions and standardised scores. The primary problem facing any study of pneumonia is accurate diagnosis. The overlap of clinical and radiological findings between severe viral infections, asthma and bacterial pneumonia can make it difficult to determine which febrile tachypneic children have wheezy diseases and which ones would benefit from antibiotic treatment. In many low-resource areas, this is further complicated by infectious diseases, such as malaria and dengue, which can have similar presentations. Early WHO tachypnea-based diagnostic protocols were intentionally over-sensitive to ensure that all children with bacterial pneumonia received antibiotics. Later attempts were made to improve the detection of wheezy diseases, by adding audible wheeze or acute bronchodilator response to the basic criteria. However, these were shown to be imprecise, particularly amongst the sickest children.

Investigators chose to formalize the diagnostic method described by Sachdev et al who classified patients into four groups (pneumonia, wheezy disease, mixed and non-respiratory) based on consultant review of a detailed history and examination plus a chest radiograph (CXR). Investigators recorded 29 items from a protocol that included history, examination, CXR and oximetry (see table). In order to combine results from data collection between centres, standardised scoring systems for conscious level and auscultation findings were used. For chest radiographs, a modification of the recently updated system recommended by the WHO was used. During the one week preparatory period, the system was explained to all involved ER physicians and pediatricians using examples and practice interpretation.

Study protocol. All children below 5 years age who present to the emergency rooms of the study hospitals with cough or difficulty breathing of less than 5 days, are identified. If their initial respiratory rate met WHO criteria for pneumonia, the study is explained by a native speaker of their primary language and they are invited to enter the study. Families are not paid to enrol but the study covers the cost of a CXR for every child plus travel expenses for outpatients to return for review on day four. After enrolment, twenty nine features of the child's history, examination and CXR are assessed by the ER physician and recorded by the study coordinator(Table 2).

After reviewing the data, the ER physician is asked to place the child into one of four diagnostic categories: pneumonia, wheezy disease (asthma and bronchiolitis), mixed (evidence of pneumonia and wheeze) and non-respiratory (malaria, dengue etc). The ER physician is solely responsible for subsequent management decisions. All study patients are reviewed four days later by a qualified pediatrician who is blinded to the ER physician's CXR interpretation and diagnosis. Based on a review of the clinical data at presentation, plus subsequent course over 4 days and a second examination, the pediatrician places the patient into one of the four diagnostic categories. This is considered the child's final diagnosis for analysis.

Statistical analysis. Logistic regression analysis will be used to determine which of the initial clinical variables had the best predictive power for pneumonia and asthma. The best cut-off values for continuous variables were established using receiver operating curve analysis. For each predictive variable, sensitivity, specificity plus positive and negative predictive value will be calculated from conventional tables using standard equations. When the predictive value of combining variables is tested, investigators will link them as 'A and/or B'. This increases sensitivity but decreases specificity, compared to using 'A and B.' Continuous variables will be displayed as mean +/- one standard deviation. Categorical variables will be displayed with box and whisker plots where the whiskers represent full range.

Table of investigations performed in the ER at presentation.

History Recorded details Cough yes/no Difficulty Breathing yes/no Lethargy yes/no Reduced feeding yes/no Fever yes/no Previous similar episodes number Vaccinations number and type

Examination Recorded details Age months Weight weight for age 'z' score Temperature ⁰ Celsius Heart rate beats/minute Respiratory rate breaths/minute Indrawing present/absent

Responsiveness score:

A fully alert V responds to voice P responds to pain U unconscious

Auscultation score:

Chest clear normal vesicular breath sounds Crackles coarse or fine inspiratory crackles/rattles Wheeze high pitched whistling noise, inspiratory or expiratory Crackles and wheeze both sounds present Bronchial breathing tracheal breath sounds heard over the lungs

Investigations Recorded details

CXR score: one or more of:

Normal ) Hyperinflation ) Minor patchy changes ) definitions, see table 3 Major patchy changes ) Lobar changes ) Pleural fluid ) Oximetry % oxygen saturation

ELIGIBILITY:
Inclusion Criteria:

* All children below 5 exceeding WHO age-dependent tachypnea criteria.

Exclusion Criteria:

* None

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study is intended to clinically relevant. All tachypneic children below 5 yrs age are eligible for enrollment. There are no exclusion criteria. Sampling will be by convenience.
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Child's diagnosis in one of four categories (pneumonia, wheezy disease, mixed and non-respiratory) | One year
  All children enrolled in the study, fulfill WHO criteria for pneumonia on day one. After assessing 29 different variables at presentation (day 1), including CXR, oximetry, pulse, respiratory rate, a qualified pediatrician makes the primary study diagnosis on day 4. Based on the results and review of progress, the consultant places the child into one of four diagnostic groups - pneumonia, wheezy disease, mixed and non-respiratory. These are the principal reference diagnoses for the rest of the analyses.

SECONDARY OUTCOMES:
Child's clinical outcome in three categories (better, worse, dead) | One year
  After diagnostic review on day 4, the child's clinical outcome is also noted. The child is placed into three outcome categories - better, worse, dead.

OTHER OUTCOMES:
Child's oxygen saturation measured by cell-phone oximeter and bedside Massimo commercial oximeter | one year
  The anesthetic department has developed a smart phone application that allows saturation readings to be made with an attachable finger probe. These readings will be compared to a those measured using a standard commercial oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Seear, FRCPC, Principal Investigator — BC's Children's Hospital
Locations (1):
- BC's Children's Hospital, Vancouver, British Columbia, Canada